CLINICAL TRIAL: NCT03853083
Title: HYPOXI for Women With Lipedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, KHerbst, Associate Professor, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1712140375
Record Dates: First submitted 2019-01-31; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxi Equipment (Experimental)
  Interventions: Device: Hypoxi Equipment
- Recumbent Bicycle (Active Comparator)
  Interventions: Device: Recumbent Bicycle

INTERVENTIONS:
Device: Hypoxi Equipment — Using the Hypoxi exercise equipment to try and improve lipedema fat tissue
  Arms: Hypoxi Equipment
Device: Recumbent Bicycle — Recumbent bike is a piece of exercise equipment used as the comparison group
  Arms: Recumbent Bicycle

SUMMARY:
The proposed study is for women with lipedema, a painful fat disorder where fat cannot be lost from the legs and hips with diet and exercise. The study will compare the use of the specialized exercise equipment called HYPOXI, which is like a bike but you lie down and air circulates around the participant's legs like a vacuum with pressure increasing and decreasing in cycles over time. The goal of the study is to see if using a HYPOXI bike compared to a regular recumbent (sit down) bike helps women with lipedema lose weight. The women with lipedema in the study will have the option to use a whole-body suit that works like a pump and was designed to improve blood circulation in the body. The body suit is called Dermology and can be used before the HYPOXI exercise equipment but will be optional for the women in the study. The study is 16 weeks long for 20 women with lipedema. Ten women with lipedema will exercise with HYPOXI for 8 weeks then switch to a recumbent bike for the second 8 weeks. The other 10 women will exercise on a recumbent bike for 8 weeks then switch to HYPOXI for 8 weeks in the second half of the study. Baseline, mid-study, and end of study data will be collected including measurements of body composition and shape, a blood draw at the beginning, middle and end, and questionnaires. This study will be listed on clinicaltrials.gov for more information.

ELIGIBILITY:
Inclusion Criteria

* Female
* 18-65 years of age
* Lipedema any stage
* Weight < 300 lbs.
* Able to participate for 4 months
* Self-reported weight stable
* Able to use Hypoxi equipment & recumbent bike
* Able to undergo baseline, mid- and end-study in Tucson.

Exclusion Criteria

* Hip width > 30 inches (76.2 cm)
* Waist width > 46 inches
* Pregnancy
* Use of weight loss medication within 3 months of the study
* History of myocardial infarction
* New York Heart Association Functional Class II or above congestive heart failure
* Sustained tachycardia above calculated maximum heart rate limit

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Bioimpedence Scale Assessment of Total Body Lean Body Mass | Change in muscle mass from baseline to end of study arm (8 weeks)
  Whole body muscle content in kilograms
Bioimpedence Scale Assessment of Total Body Fat Mass | Change in fat mass from baseline to end of study arm (8 weeks)
  Whole body fat mass in kilograms
Bioimpedence Scale Assessment of Total Body Water | Change in total body water from baseline to end of study arm (8 weeks)
  Total body water in kilograms

SECONDARY OUTCOMES:
Resting energy expenditure | Change in resting energy expenditure from baseline to end of study arm (8 weeks)
  Resting energy expenditure by MedGem Device in kcal/day
Waist/Hip ratio | Change in waist/hip ratio from baseline to end of study arm (8 weeks)
  Waist and hip measurements using a tape measure; this is a ratio with no units